CLINICAL TRIAL: NCT02280876
Title: Randomized, Comparative, Double Blind Controlled Phase II Clinical Trial, to Evaluate the Efficacy of ApE in Patients With Multiple Sclerosis (MS).
Brief Title: Efficacy Study of Andrographis Paniculata Purified Standardized Extract (ApE) in Patients With Multiple Sclerosis (MS)
Acronym: PCNS-EM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidad Austral de Chile (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government); University of Chile (Other)
Responsible Party: Principal Investigator, Juan C. Bertoglio, MD, Principal Clinical Investigator, Universidad Austral de Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PaCRU-02/PCNS.EM/12; PCNS-EM (Other Grant/Funding Number: FONDEF D09I1085 (CONICYT - Chile))
Record Dates: First submitted 2014-10-20; First posted 2014-11-03 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: MS; Demyelinating Autoimmune Diseases; CNS; Nervous System Diseases
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Nervous System Diseases | interventions — andrographolide; Andrographis paniculata extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 - Andrographis paniculata p/st extract (Active Comparator): 1 - Andrographis paniculata extract. Active comparator, consists of 15 adult patients with active Recurrent Remitting Multiple Sclerosis, randomly assigned, taking the active test product (Andrographis paniculata p/st extract, oral lozenges, one BID, for 12 months), in addition to base medication (Interferon).
  Interventions: Drug: 1 - Andrographis paniculata p/st extract
- 2 - Excipients (Placebo Comparator): 2 - Excipients. Placebo comparator, consists of 15 adult patients with active Recurrent Remitting Multiple Sclerosis, randomly assigned, taking the placebo formulation (Only the excipients of the active test product, in oral lozenges of same shape, one BID, for 12 months), in addition to base medication (Interferon).
  Interventions: Drug: 2 - Excipients

INTERVENTIONS:
Drug: 1 - Andrographis paniculata p/st extract — Andrographis paniculata Extract (ApE), Oral tablets 650 mg, with 170 mg. of andrographolides active principles, three times per day, during a total of 365 continuous days.
  Other Names:
  • ApE tablets, EUROMED Specific. Santiago Chile.
  Other Names: Andrographolide; Verum formulation; Andrographis paniculata Extract ( ApE ); Paractin®
  Arms: 1 - Andrographis paniculata p/st extract
Drug: 2 - Excipients — Placebo 650mg tabs, 2/day, 365 days continuously.
  Other Names:
  • Excipients tablets EUROMED Specific. Santiago Chile
  Other Names: Placebo formulation
  Arms: 2 - Excipients

SUMMARY:
To evaluate the efficacy of ApE coated tablets, on the relapse rate in a group of relapsing remitting multiple sclerosis (RRMS) patients, as compared to a placebo group in a period of 12 months. This study will also determine the safety and tolerability of the drug administered over interferon beta vs. administration of a placebo formulation (also over interferon) during the evaluation period. Response will be assessed and measured by daily self patient recording, monthly clinical neurologist, and every three months serological and magnetic resonance parameters.

Place of Study: National study in Chile with one center at the Regional Hospital in the city of Valdivia, including 30 patients enrolled by their respective neurologists.

DETAILED DESCRIPTION:
Introduction: Multiple sclerosis is a chronic inflammatory demyelinating disease of the central nervous system that predominantly affects young adults (1). Although its etiology has not yet been elucidated, evidence points to an autoimmune pathogenesis where it is thought that self-reactive and myelin-specific cluster of differentiation four and eight (CD4)and (CD8) T cells, play an important role by reacting and destroying the myelin sheath (2). No plasma biomarkers to determine disease activity by routine clinical measurements, the existence a pattern of pro-inflammatory cytokines has been described, with range increased Interferon (IFN), Tumoral Necrosis Factor alpha (TNFa) and Interleukin 12 (IL-12), as well as a decline in Interleukin10 (IL10) and Interleukin 4 (IL4) anti-inflammatory cytokines (3). To date, the most common treatment for MS is Interferon beta immunomodulation, although its cost / effectiveness has been questioned4.

Regardless of the progressive form and the existence of outbreaks, the fatigue symptom is one of the most frequent and disabling one in patients with MS. The proposed pathogenic mechanisms are multiple, although its exact pathophysiology is unknown. Also, there is still no treatment that has proven to be completely effective in stopping the progression of the disease (5). Description of the botanical drug to be used in this clinical research: The botanical drug to be used in this clinical research, is a phytopharmaceutical tablet made by Good Manufacturing Practices (GMP) containing a purified, standardized and patented extract of Andrographis paniculata Nees (Acanthaceae) {U.S. Patent: 8,084,495 B2; Date: Dec. 27, 2011} (ApE).

This is a medicinal annual plant, native to India and China whose active compounds are bitter diterpenoid lactones such as and especially 14-deoxyandrographolide, Neoandrographolide and specially Andrographolide, which has proven particularly effective in regulating the immune response (7, 9).

The cellular and molecular mechanisms responsible for the immunomodulatory and anti-inflammatory properties of Andrographolide, are for the most part still unknown. However, recent studies with in vitro and in vivo assays indicate that 10 micromol (µM) per liter inhibits Tumoral Necrosis Factor Beta (NF-kB). Specifically, Andrographolide at concentrations of 10 micromol (uM) per liter interferes with DNA binding of NF-kB (10), by reducing the expression of COX-2 in neutrophils induced with Formyl-Methionyl-Leucyl-Phenylalanine (fMLP) and Platelet Activating Factor (PAF). Moreover, Andrographolide reduces Interferon gamma (IFNg) and IL-2 production in Concanavalin A (Con A) induced T-cells, without affecting cell viability or inducing apoptosis, also diminishing thymocyte apoptosis induced by corticosteroids. Furthermore, Andrographolide and 14-deoxyandrographolide are capable of inhibiting extracellular signal-regulated kinases 1/2 (ERK1/2) phosphorylation in T cells and neutrophils, respectively (11, 12).

Security settings: Toxicity and Tolerance Analysis of acute and sub-chronic toxicity of ApE in rodents and pigs, using the basic component of ApE have been carried out in our laboratory at the Institute of Pharmacology and Toxicology, Universidad Austral de Chile, and according to the guidelines of Good Laboratory Practice (GLP) of the Food Administration Agency (FDA). Also, clinical phase I and II clinical studies have been performed, plus controlled daily treatment of 12 patients with different rheumatoid conditions and other 8 patients with Recurrent Remitting Multiple Sclerosis (RRMS) for more than five years. All these observations have proven a wide range of dosage safety without any detected toxic effects at therapeutic dose of 2 milligrams per kilogram of body weight.

Hypothesis: In experimental inflammatory and human autoimmune diseases, such as Rheumatoid arthritis and related conditions (17, 19), and also in animal models in which Experimental Autoimmune Encephalitis (EAE) is induced, we have recently shown that Andrographolide can significantly reduce the clinical symptoms and outcome of this diseases (6), for which we have now proposed this clinical study in RRMS.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with MS according to McDonald scale
* Relapsing Remitting Forms of MS (subtypes of Lublin)
* Minor or less incapacity according to EDSS scale
* At least one relapse in the last 2 years
* Sign an informed consent

Exclusion Criteria:

* Primary and Secondary Progressive MS patients.
* Use of corticosteroids up to one month previous to enrollment
* Use of immunosuppressors up to one month previous to enrollment
* Use of drugs that induce hepatic metabolism
* Pregnancy, contraception, breast feeding.
* Psychiatric disorders
* Systemic diseases
* Chronic renal failure
* Diabetes mellitus
* Cardiac failure
* Respiratory failure
* Cancer

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Clinical inflammatory (stamina) and disability score parameters (sensorial, neurosensitive, neuromotor and cognitive function) in patients with RRMS, treated with ApE and placebo administered over beta interferon. | 12 months
  Clinical parameters (stamina, sensorial, neurosensitive, neuromotor and cognitive function), will be measured by the Fatigue Severity Scale (FSS) and Expanded Disability Scale (EDSS) in patients with RRMS treated with ApE and placebo.

SECONDARY OUTCOMES:
Safety, tolerability and efficacy of ApE and placebo administered over beta interferon in RRMS treated patients (adverse symptoms, general clinical laboratory and comparative statistical parameters) | 12 months
  Patients dairy of possible adverse symptoms, general clinical laboratory and comparative statistical parameters

OTHER OUTCOMES:
Central Nervous System (CNS) local inflammatory activity and anatomical damage parameters (functional and structural lesions) in RRMS patients treated with ApE and placebo administered over beta interferon. | 12 months
  CNS number, size, location and gadolinium uptaking of lesions in brain and / or spine will be measured by magnetic resonance (MR) at 0, 3, 6 and 12 months.
Plasmatic inflammatory activity parameters (cytokines) in RRMS patients treated with ApE and placebo administered over beta interferon. | 12 months
  Plasmatic levels of IFNg, Interleukin 17 (IL17), Interleukin IL10, Interleukin 6 (IL6), IL4, TNFa, will be measured at 0, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Juan L. Hancke, PhD, Study Director — Universidad Austral de Chile
Locations (1):
- Hospital Regional, Valdivia, Los Ríos Region, Chile

IPD SHARING:
Plan to Share IPD: Yes
All these trial results, will be submitted to publication in a major journal of the specialty, upon conclusion of data processing and evaluation.

REFERENCES:
- [Background] Noseworthy JH, Lucchinetti C, Rodriguez M, Weinshenker BG. Multiple sclerosis. N Engl J Med. 2000 Sep 28;343(13):938-52. doi: 10.1056/NEJM200009283431307. No abstract available. PMID 11006371
- [Background] Wingerchuk DM, Lucchinetti CF, Noseworthy JH. Multiple sclerosis: current pathophysiological concepts. Lab Invest. 2001 Mar;81(3):263-81. doi: 10.1038/labinvest.3780235. PMID 11310820
- [Background] Galboiz Y, Miller A. Immunological indicators of disease activity and prognosis in multiple sclerosis. Curr Opin Neurol. 2002 Jun;15(3):233-7. doi: 10.1097/00019052-200206000-00002. PMID 12045718
- [Background] Phillips JT, Rice G, Frohman E, Vande Gaer L, Scott T, Haas J, Eggenberger E, Freedman MS, Stuart W, Cunha L, Jacobs L, Oger J, Arnold D, Murray TJ, DiBiase M, Jethwa V, Goelz S. A multicenter, open-label, phase II study of the immunogenicity and safety of a new prefilled syringe (liquid) formulation of Avonex in patients with multiple sclerosis. Clin Ther. 2004 Apr;26(4):511-21. doi: 10.1016/s0149-2918(04)90053-7. PMID 15189748
- [Background] Iruretagoyena MI, Tobar JA, Gonzalez PA, Sepulveda SE, Figueroa CA, Burgos RA, Hancke JL, Kalergis AM. Andrographolide interferes with T cell activation and reduces experimental autoimmune encephalomyelitis in the mouse. J Pharmacol Exp Ther. 2005 Jan;312(1):366-72. doi: 10.1124/jpet.104.072512. Epub 2004 Aug 26. PMID 15331658
- [Background] Rajagopal S, Kumar RA, Deevi DS, Satyanarayana C, Rajagopalan R. Andrographolide, a potential cancer therapeutic agent isolated from Andrographis paniculata. J Exp Ther Oncol. 2003 May-Jun;3(3):147-58. doi: 10.1046/j.1359-4117.2003.01090.x. PMID 14641821
- [Background] Calabrese C, Berman SH, Babish JG, Ma X, Shinto L, Dorr M, Wells K, Wenner CA, Standish LJ. A phase I trial of andrographolide in HIV positive patients and normal volunteers. Phytother Res. 2000 Aug;14(5):333-8. doi: 10.1002/1099-1573(200008)14:53.0.co;2-d. PMID 10925397
- [Background] Hidalgo MA, Romero A, Figueroa J, Cortes P, Concha II, Hancke JL, Burgos RA. Andrographolide interferes with binding of nuclear factor-kappaB to DNA in HL-60-derived neutrophilic cells. Br J Pharmacol. 2005 Mar;144(5):680-6. doi: 10.1038/sj.bjp.0706105. PMID 15678086
- [Background] Burgos RA, Hidalgo MA, Monsalve J, LaBranche TP, Eyre P, Hancke JL. 14-deoxyandrographolide as a platelet activating factor antagonist in bovine neutrophils. Planta Med. 2005 Jul;71(7):604-8. doi: 10.1055/s-2005-871264. PMID 16041644
- [Background] Burgos RA, Seguel K, Perez M, Meneses A, Ortega M, Guarda MI, Loaiza A, Hancke JL. Andrographolide inhibits IFN-gamma and IL-2 cytokine production and protects against cell apoptosis. Planta Med. 2005 May;71(5):429-34. doi: 10.1055/s-2005-864138. PMID 15931581
- [Background] Coon JT, Ernst E. Andrographis paniculata in the treatment of upper respiratory tract infections: a systematic review of safety and efficacy. Planta Med. 2004 Apr;70(4):293-8. doi: 10.1055/s-2004-818938. PMID 15095142
- [Background] Thamlikitkul V, Dechatiwongse T, Theerapong S, Chantrakul C, Boonroj P, Punkrut W, Ekpalakorn W, Boontaeng N, Taechaiya S, Petcharoen S, et al. Efficacy of Andrographis paniculata, Nees for pharyngotonsillitis in adults. J Med Assoc Thai. 1991 Oct;74(10):437-42. PMID 1797953
- [Background] Caceres DD, Hancke JL, Burgos RA, Wikman GK. Prevention of common colds with Andrographis paniculata dried extract. A Pilot double blind trial. Phytomedicine. 1997 Jun;4(2):101-4. doi: 10.1016/S0944-7113(97)80051-7. PMID 23195395
- [Background] Cabrera D, Gutierrez J, Cabello-Verrugio C, Morales MG, Mezzano S, Fadic R, Casar JC, Hancke JL, Brandan E. Andrographolide attenuates skeletal muscle dystrophy in mdx mice and increases efficiency of cell therapy by reducing fibrosis. Skelet Muscle. 2014 Mar 21;4:6. doi: 10.1186/2044-5040-4-6. eCollection 2014. PMID 24655808
- [Background] Caceres DD, Hancke JL, Burgos RA, Sandberg F, Wikman GK. Use of visual analogue scale measurements (VAS) to asses the effectiveness of standardized Andrographis paniculata extract SHA-10 in reducing the symptoms of common cold. A randomized double blind-placebo study. Phytomedicine. 1999 Oct;6(4):217-23. doi: 10.1016/S0944-7113(99)80012-9. PMID 10589439
- [Background] Gabrielian ES, Shukarian AK, Goukasova GI, Chandanian GL, Panossian AG, Wikman G, Wagner H. A double blind, placebo-controlled study of Andrographis paniculata fixed combination Kan Jang in the treatment of acute upper respiratory tract infections including sinusitis. Phytomedicine. 2002 Oct;9(7):589-97. doi: 10.1078/094471102321616391. PMID 12487322
- [Background] Burgos RA, Hancke JL, Bertoglio JC, Aguirre V, Arriagada S, Calvo M, Caceres DD. Efficacy of an Andrographis paniculata composition for the relief of rheumatoid arthritis symptoms: a prospective randomized placebo-controlled trial. Clin Rheumatol. 2009 Aug;28(8):931-46. doi: 10.1007/s10067-009-1180-5. Epub 2009 Apr 29. PMID 19408036
- [Result] Bertoglio JC, Baumgartner M, Palma R, Ciampi E, Carcamo C, Caceres DD, Acosta-Jamett G, Hancke JL, Burgos RA. Andrographis paniculata decreases fatigue in patients with relapsing-remitting multiple sclerosis: a 12-month double-blind placebo-controlled pilot study. BMC Neurol. 2016 May 23;16:77. doi: 10.1186/s12883-016-0595-2. PMID 27215274
- See also: María A. Hidalgo, Juan L. Hancke, Juan C. Bertoglio and Rafael A. Burgos. Andrographolide, a New Potential Drug for the Long Term Treatment of Rheumatoid Arthritis Disease. Innovative Rheumatology. International standard book (ISBN) 978-953-51-0916-7 — http://www.intechopen.com/books/innovative-rheumatology/andrographolide-a-new-potential-drug-for-the-long-term-treatment-of-rheumatoid-arthritis-disease